CLINICAL TRIAL: NCT03956576
Title: Apelin as a Potential Treatment for Chronic Kidney Disease: The AlPaCKa Study
Brief Title: Apelin as a Potential Treatment for Chronic Kidney Disease
Acronym: AlPaCKa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Kidney Cancer UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AC18094
Record Dates: First submitted 2018-12-11; First posted 2019-05-20 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Chronic Kidney Diseases; Cardiovascular Diseases; Endothelial Dysfunction
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases | interventions — apelin 13, Pyr(1)-

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic Kidney Disease patients (Active Comparator): Forearm blood flow studies
  - acetylcholine (7.5, 15, 30microgram/min), sodium nitroprusside (1, 2, 4microgram/min) and [Pyr1]apelin-13 (0.3, 1, 3, 10, 30, 100nmol/min). Incremental doses of each lasting 8 minutes with saline washout between drugs.
  Renal clearance studies
  * Two standard para-aminohippurate (PAH) / iohexol clearance studies with infusion of either apelin or placebo on each day.
  * Dose of PAH / iohexol dependent on renal function. Continuous infusion lasting 6.5hours in total.
  * [[Pyr1]apelin-13 infusions: 1nmol/min and 30nmol/min for 30 minutes each.
  Interventions: Other: [Pyr]apelin-13
- Healthy volunteers (Active Comparator): Forearm blood flow studies
  - acetylcholine (7.5, 15, 30microgram/min), sodium nitroprusside (1, 2, 4microgram/min) and [Pyr1]apelin-13 (0.3, 1, 3, 10, 30, 100nmol/min). Incremental doses of each lasting 8 minutes with saline washout between drugs.
  Renal clearance studies
  * Two standard para-aminohippurate (PAH) / iohexol clearance studies with infusion of either apelin or placebo on each day.
  * Dose of PAH / iohexol dependent on renal function. Continuous infusion lasting 6.5hours in total.
  * [Pyr1]apelin-13 infusions: 1nmol/min and 30nmol/min for 30 minutes each.
  Interventions: Other: [Pyr]apelin-13

INTERVENTIONS:
Other: [Pyr]apelin-13 — Peptide [Pyr]apelin-13 infusion

SUMMARY:
Chronic kidney disease (CKD) affects 8-16% of the world's population, and is independently associated with cardiovascular disease (CVD). As renal function declines, rates of major adverse cardiovascular events, cardiovascular and all-cause mortality increase. In addition to hypertension, increased arterial stiffness is characteristic of CKD, a marker of CVD risk, and an independent predictor of mortality in CKD patients. The endothelium is an important regulator of arterial stiffness, and endothelial dysfunction is a feature of CKD and a predictor of CVD. Current treatment of CKD is limited and aims to reduce blood pressure and proteinuria through the use of angiotensin converting enzyme (ACE) inhibitors or angiotensin receptor blockers (ARB). However, many patients still progress to end-stage renal failure and often these patients die as a result of CVD.

A novel peptide, apelin, is proposed to be a potential treatment for CKD, with additional cardiovascular benefits. The AlPaCKa study investigators will carry out forearm blood flow and renal clearance studies in 25 patients with CKD and 25 matched healthy volunteers to determine the effects of apelin on cardiovascular and renal parameters. It is hoped apelin will be confirmed as a potential future treatment for CKD.

DETAILED DESCRIPTION:
The apelins are a family of peptides whose most abundant isoform is [Pyr1]apelin-13. This binds to a single G protein coupled receptor known as 'APJ', which is widely expressed particularly in endothelium and cardiomyocytes. Apelin is the most powerful inotropic agent discovered to date, and apelin infusion into healthy humans leads to endothelium-dependent vasodilatation and BP lowering. Given its vasodilatory and inotropic effects, apelin is being investigated as a novel therapy for heart failure and pulmonary arterial hypertension, both of which are features of CKD. The apelin/APJ system is widely expressed in the human kidney (endothelium, smooth muscle cells, glomeruli) with a predominance in the renal medulla. It is recognised to have a role in fluid homeostasis, and apelin infusion in rodents leads to a dose-dependent diuresis but it is difficult to discriminate how much of this is due to renal vasodilatation as opposed to a direct tubular effect. However, it has been shown that apelin counteracts the antidiuretic effect of vasopressin at the tubular level. Evidence therefore suggests that apelin could have additional cardioprotective effects in CKD and could promote natriuresis and diuresis. To date there are no clinical studies of the actions of apelin in the kidney in health or CKD, or its effect on systemic haemodynamics in CKD.

Twenty-five patients with CKD and 25 matched healthy volunteers will undergo forearm blood flow studies with acetylcholine, sodium nitroprusside and apelin to determine the local haemodynamic effects of apelin in CKD, specifically the effects on endothelial function. The same subjects will then complete two renal clearance studies during systemic apelin / placebo infusion (randomised and double-blinded), by standard renal para-aminohippurate and inulin clearance techniques. Blood and urine samples will be collected every 30 minutes. This will allow the effects of apelin on renal function, renal blood flow, proteinuria, natriuresis and diuresis to be demonstrated. Cardiovascular effects will be determined by systemic bioimpedance measures and pulse wave velocity. This study aims to open a new area of clinical research with apelin.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18yrs
* Stable, non-diabetic chronic kidney disease stages 1 - 4 as defined by Kidney Disease: Improving Global Outcomes (KDIGO) 2012 classification (estimated Glomerular Filtration Rate (eGFR) >15ml/min/1.73m2)
* Clinically optimised on an angiotensin converting enzyme inhibitor / angiotensin receptor blocker, or intolerant to these agents.

Exclusion Criteria:

* Age <18 years
* Diabetes mellitus
* Overt cardiovascular disease
* Blood pressure >160/100mmHg
* Estimated GFR of <15ml/min/1.73m2
* Renal transplant recipients
* Haemodialysis / peritoneal dialysis patients
* Serum albumin <30g/L
* Patients receiving tolvaptan therapy for polycystic kidney disease
* Patients not medically fit to attend for study visits
* Patients without mental capacity or willingness to provide informed consent
* History of multiple and/or severe allergic reaction to drugs (including study drugs) or food
* Patients who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Change in forearm blood flow | 1 hour
  Venous occlusion plethysmography
Change in renal blood flow | 4 hours
  Para-aminohippurate clearance study

SECONDARY OUTCOMES:
Change in arterial stiffness | 1 hour
  Pulse wave velocity measures
Change in natriuresis | 4 hours
  Urinary sodium excretion measures
Change in diuresis | 4 hours
  Free water clearance measurement
Change in blood pressure | 4 hours
  Blood pressure monitoring
Change in proteinuria | 4 hours
  Urinary protein excretion
Change in chorioretinal metrics as assessed by optical coherence tomography (OCT | 4 hours
  Optical coherence tomography measurements

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Dhaun, PhD, Principal Investigator — University of Edinburgh
Locations (1):
- Clinical Research Centre, Western General Hospital, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No data to be shared

REFERENCES:
- [Derived] Chapman FA, Melville V, Godden E, Morrison B, Bruce L, Maguire JJ, Davenport AP, Newby DE, Dhaun N. Cardiovascular and renal effects of apelin in chronic kidney disease: a randomised, double-blind, placebo-controlled, crossover study. Nat Commun. 2024 Oct 14;15(1):8387. doi: 10.1038/s41467-024-52447-7. PMID 39402039